CLINICAL TRIAL: NCT05184062
Title: A Phase II Double-blind, Placebo-controlled Study to Evaluate the Safety and Tolerability of AZD7442 in Chinese Adults
Brief Title: A Study to Evaluate the Safety and Tolerability of AZD7442 in Chinese Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: D8850C00008
Record Dates: First submitted 2021-11-17; First posted 2022-01-11 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-09

CONDITIONS: Coronavirus Disease 2019 (COVID-19)
Keywords: Coronavirus; COVID-19; AZD7442
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — cilgavimab and tixagevimab drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AZD7442 (Experimental): co-administration of a single dose of 600 mg AZD7442 (300 mg AZD8895 and 300 mg AZD1061) by intravenous (IV) infusion.
  Interventions: Drug: 600 mg AZD7442 IV
- Placebo (Placebo Comparator): co-administration of a single dose of 600mg placebo by intravenous (IV) infusion.
  Interventions: Drug: 600mg placebo IV

INTERVENTIONS:
Drug: 600 mg AZD7442 IV — Participants will be randomized to receive co-administration of 600 mg AZD7442 (300 mg AZD8895 and 300 mg AZD1061) by a single IV infusion.
  Other Names: AZD7442
  Arms: AZD7442
Drug: 600mg placebo IV — Participants will be randomized to receive co-administration of 600mg placebo by a single IV infusion.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
To evaluate the safety and tolerability of a single dose of 600 mg AZD7442 administered IV (intravenous) to Chinese adults (including those with stable medical conditions).

DETAILED DESCRIPTION:
A Phase II, randomised, double-blind, placebo-controlled study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of AZD7442 for administration to prevent and treat coronavirus disease 2019 (COVID-19) in Chinese adult participants (including healthy participants as well as participants with stable medical conditions), approximately 479 days in duration for each participant.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years
2. Negative results of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) quantitative reverse transcriptase polymerase chain reaction (qRT-PCR)
3. Healthy or medically stable participants
4. Contraceptive within 365 days post dosing

Exclusion Criteria:

1. Medical condition:

   * Known hypersensitivity to monoclonal antibody (mAb) or investigational product (IP) component.
   * Acute illness including fever on the day prior to or day of dosing.
   * Any other significant disease increase the risk to participant study.
2. Laboratory related:

   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.0 × upper limit of normal (ULN), alkaline phosphatase (ALP) > 1.5 × ULN, or TBL (total bilirubin) > 1.5 × ULN (unless due to Gilbert's syndrome).
   * Serum creatinine > 176 μmol/L.
   * Haemoglobin < 10g/dL.
   * Platelet count < 100 × 10^3/μL.
   * White blood cell count < 3.5 × 10^3/μL or neutrophil count < 1.5 × 10^3/μL.
   * Other laboratory significantly abnormal in the screening panel that, in the opinion of the investigator, will increase participants risk or might confound analysis of study results.
3. COVID-19 infection history/any receipt of mAb indicated for COVID-19.
4. Prior/concomitant treatment: Receipt of any investigational product within 90 days or 5 antibody half-lives (whichever is longer) prior to Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2023-05-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Research Site, Baoding
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Lanzhou
  - Research Site, Shanghai
  - Research Site, Suzhou
  - Research Site, Ürümqi
  - Research Site, Xuzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Zhang J, Zhang H, Zhang Y, Liu S, Ge X, Zhang H, Li Y, Chen CC, Stepanov O, Tang W, Zhang W. Safety and Pharmacokinetics of Long-Acting Monoclonal Antibodies Tixagevimab and Cilgavimab (AZD7442) in a China Phase 2 Study and Evaluation of Asian Race Effect. Clin Pharmacol Drug Dev. 2025 Nov;14(11):846-855. doi: 10.1002/cpdd.1586. Epub 2025 Sep 5. PMID 40910575
- [Derived] Hirsch C, Park YS, Piechotta V, Chai KL, Estcourt LJ, Monsef I, Salomon S, Wood EM, So-Osman C, McQuilten Z, Spinner CD, Malin JJ, Stegemann M, Skoetz N, Kreuzberger N. SARS-CoV-2-neutralising monoclonal antibodies to prevent COVID-19. Cochrane Database Syst Rev. 2022 Jun 17;6(6):CD014945. doi: 10.1002/14651858.CD014945.pub2. PMID 35713300
- See also: CSR_synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8850C00008&attachmentIdentifier=43f718b5-e390-4747-88ec-be54e7c3d61d&fileName=d8850c00008-study-synopsis_pLSLV_Redacted.pdf&versionIdentifier=
- See also: protocol_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8850C00008&attachmentIdentifier=96ccfa2e-8ac7-416c-9643-c13074e28928&fileName=d8850c00008-csp-v2_Redacted.pdf&versionIdentifier=
- See also: SAP_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8850C00008&attachmentIdentifier=77761e0e-2fae-4593-b09e-27161cb00ee3&fileName=d8850c00008-sap-ed-2_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- AZD7442: AZD7442 600 mg IV
- Placebo: Placebo Group
Period: Overall Study
Arm/Group | AZD7442 | Placebo
Started | 202 (The study consists of 3 periods: Screening period: Days -28 through -1 (up to 28 days), Intervention period: Day 1, randomisation and dosing, Safety follow-up period: Days 2 through 451 (450 days).) | 70
Completed | 196 | 69
Not Completed | 6 | 1
Not completed — Lost to Follow-up | 5 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD7442 | Placebo | Total
Number analyzed (Participants) | 202 | 70 | 272
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.67 (11.73) | 35.71 (12.05) | 34.2 (11.80)
Age, Customized [Number; unit: Participants]
  >60 years | 12 | 4 | 16
  18 - 44 years | 170 | 54 | 224
  45 -60 years | 20 | 12 | 32
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Safety Analysis Set
  Participants
    Female | 62 | 22 | 84
    Male | 140 | 48 | 188
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 202 | 70 | 272
Race/Ethnicity, Customized [Number; unit: Participants]
  Not Hispanic or Latino | 202 | 70 | 272
COVID-19 vaccination status [Count of Participants; unit: Participants]
  No, non-vaccinated | 98 | 34 | 132
  Yes, vaccinated | 104 | 36 | 140
Baseline Weight [Mean (Standard Deviation); unit: kg] | 67.26 (11.54) | 66.51 (9.91) | 67.07 (11.13)
Baseline Height [Mean (Standard Deviation); unit: cm] | 167.50 (8.77) | 166.53 (7.78) | 167.25 (8.53)
Baseline Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 23.84 (3.14) | 23.91 (2.96) | 23.86 (3.09)

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events of Special Interest
Description: Adverse events of special interest are events of scientific and medical interest, specific to the further understanding of the study intervention safety profile, and require close monitoring and rapid communication by the investigators to the sponsor.
Time Frame: recorded from the time of signature of the ICF up to 245 days
Measure: Count of Participants; unit: Participants
Arm/Group | AZD7442 | Placebo
Number analyzed (Participants) | 202 | 70
Participants | 0 | 0

2. Secondary Outcome: Serum Concentrations of AZD7442 Over Time
Description: Serum concentrations for each scheduled time point are summarized based on the PK Analyses Set using descriptive statistics
Time Frame: recorded from the time of signature of the ICF through the last participant contact. Protocol-specified timepoints include Pre-dose, Day 1, Day 8, Day 31, Day 61, Day 91, Day 181, Day 271, and Day 361.
Population: All participants who received AZD7442 and had at least one quantifiable serum PK observation post-dose, with no important protocol deviations thought to impact the analysis of the PK data
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | AZD7442
Number analyzed (Participants) | 202
μg/mL
  pre-dose | 0 (0)
  Day 1 | 219.7 (37.81)
  Day 8 | 136.1 (26.58)
  Day 31 | 101.5 (19.99)
  Day 61 | 74.60 (16.08)
  Day 91 | 55.98 (12.82)
  Day 181 | 28.92 (7.752)
  Day 271 | 12.74 (4.186)
  Day 361 | 5.858 (2.530)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time of signature of the informed consent form up to 445 days.
Arm/Group | AZD7442 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/202 | 0/70
Serious Adverse Events (participants affected / at risk) | 6/202 | 3/70
Other Adverse Events (participants affected / at risk) | 144/202 | 58/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD7442 (N=202) | Placebo (N=70)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Laryngopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD7442 (N=202) | Placebo (N=70)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menstruation delayed (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (4)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 3 (3) | 0 (0)
Lip blister (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 2 (2) | 0 (0)
Noninfective gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 3 (3) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Discomfort (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2)
Infusion site oedema (General disorders) | 1 (1) | 0 (0)
Infusion site swelling (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 7 (7) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Nodal rhythm (Cardiac disorders) | 2 (2) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 1 (2) | 0 (0)
Cervicitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 3 (3) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 4 (4)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Pericoronitis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1)
Otolithiasis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Tinea cruris (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 29 (36) | 13 (15)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Mouth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 8 (8) | 3 (3)
Blood glucose increased (Investigations) | 4 (7) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Blood pressure increased (Investigations) | 2 (6) | 0 (0)
Blood urine present (Investigations) | 1 (1) | 1 (1)
C-reactive protein increased (Investigations) | 4 (4) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 3 (4) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Monocyte count increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 2 (2)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 0 (0)
Protein urine present (Investigations) | 15 (17) | 9 (10)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2) | 0 (0)
Qrs axis abnormal (Investigations) | 1 (1) | 0 (0)
Bile acids increased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 3 (3)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyperphagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 4 (4)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Albuminuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (3) | 2 (2)
Proteinuria (Renal and urinary disorders) | 2 (3) | 0 (0)
Urine abnormality (Renal and urinary disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cystic lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Seborrhoeic alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 20 (20) | 4 (4)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic calcification (Hepatobiliary disorders) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 58 (58) | 20 (20)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Infection parasitic (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 12 (12) | 14 (14)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 1 (1)
Myocardial necrosis marker increased (Investigations) | 0 (0) | 1 (1)
Ultrasound liver abnormal (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Red blood cell count decreased (Investigations) | 0 (0) | 1 (1)
White blood cells urine positive (Investigations) | 1 (1) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Type V hyperlipidaemia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hyperadrenocorticism (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Alcohol use (Social circumstances) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-08-27): https://cdn.clinicaltrials.gov/large-docs/62/NCT05184062/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT05184062/SAP_001.pdf